CLINICAL TRIAL: NCT02905279
Title: Enhancing Exposure Therapy for Spider Phobia With the Use of Threat-Relevant and Threat-Irrelevant Opposite Actions
Brief Title: Spider Phobia Opposite Action Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Doctoral student running the study left for internship and did not finish the study
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-07-0020
Record Dates: First submitted 2016-08-23; First posted 2016-09-19 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Specific Phobia
Keywords: spider phobia; animal phobia; exposure therapy; biofeedback; relaxation training
MeSH Terms: conditions — Phobia, Specific; Arachnophobia; Zoophobia | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Biofeedback (Active Comparator): Biofeedback Relaxation Training
  Interventions: Behavioral: Biofeedback Relaxation Training
- Standard Exposure (Active Comparator): Exposure Therapy
  Interventions: Behavioral: Exposure Therapy
- Exposure with Threat-Relevant OAs. (Experimental): Exposure with Threat-Relevant Opposite Actions
  Interventions: Behavioral: Exposure with Threat-Relevant Opposite Actions
- Exposure with Threat-Irrelevant OAs (Experimental): Exposure with Threat-Irrelevant Opposite Actions
  Interventions: Behavioral: Exposure with Threat-Irrelevant Opposite Actions

INTERVENTIONS:
Behavioral: Biofeedback Relaxation Training — Participants will receive one-session biofeedback relaxation training (24 minutes) for anxiety reduction. Prior to biofeedback, participants will receive education about spiders and the development and maintenance of spider phobia.
  Arms: Biofeedback
Behavioral: Exposure Therapy — Participants will receive one-session exposure therapy (24 minutes) for fear of spiders. Prior to exposure therapy, participants will receive education about spiders and the development and the development and maintenance of spider phobia.
  Arms: Standard Exposure
Behavioral: Exposure with Threat-Relevant Opposite Actions — Participants will receive one-session exposure therapy (24 minutes) for fear of spiders. During exposure, participants will engage in actions opposite to the tendencies associated with threat avoidance. Prior to exposure therapy, participants will receive education about spiders and the development and maintenance of spider phobia.
  Arms: Exposure with Threat-Relevant OAs.
Behavioral: Exposure with Threat-Irrelevant Opposite Actions — Participants will receive one-session exposure therapy (24 minutes) for fear of spiders. During exposure therapy, participants will engage in actions opposite of the action tendencies associated with the fear, but unrelated to the specific threats associated with spider phobia. Prior to exposure therapy, participants will receive education about spiders and the development and maintenance of spider phobia.
  Arms: Exposure with Threat-Irrelevant OAs

SUMMARY:
This study tests the effectiveness of exposure therapy for fear of spiders as enhanced by the use of antagonistic or opposite actions during treatment. The goal of the study is to compare the efficacy threat-relevant opposite actions and threat-irrelevant opposite actions in extinguishing fear.

DETAILED DESCRIPTION:
This study tests whether exposure therapy for fear of spiders can be enhanced with the use of opposite actions, which are actions opposite to fear-related action tendencies. The investigators will test two sub-types of opposite actions (a) threat-relevant opposite actions, which are actions antagonistic to specific threats associated with spider phobia, and (b) threat-irrelevant opposite actions, which are actions antagonistic to the fear response, but unrelated to specific threats associated with spider phobia. This exposure therapy enhanced with opposite actions will be compared with two control groups: standard exposure therapy and non-specific anxiety treatment (biofeedback relaxation training).

Individuals between the ages of 18-65 with elevated fear of spiders are randomly assigned to one of four treatment conditions (1) biofeedback relaxation training, (2) standard exposure therapy, (3) exposure therapy with threat-relevant opposite actions, and (4) exposure therapy with threat-irrelevant opposite actions. All participants undergo an online prescreen and a face-to-face screening assessment to determine eligibility and baseline (pre-treatment) symptom severity. Participants additionally complete assessments directly after treatment (post-treatment), and approximately two weeks after treatment (follow-up). The pre-treatment assessment occurs on the same day as treatment, the post-treatment assessment occurs during the treatment visit as soon as the treatment procedure is complete, and the follow-up assessment occurs within a window of 14-21 days after the completion of treatment. Participants complete two behavioral approach tests (in the treatment context and in the generalization context) at pre-treatment, post-treatment, and follow-up. Participants complete a battery of self-report questionnaires at pre-treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At Prescreen:

  * Total score of greater than or equal to 70 on the Fear of Spiders - Questionnaire (with higher scores indicating higher fear levels).
  * Indicates ongoing fear of spiders and inability to complete close approach towards spiders on brief questionnaire.
* At Screening visit: inability to complete close approach toward spiders as determined by the treatment context and generalization context Behavioral Approach Tests

Exclusion Criteria:

* Currently receiving psychotherapy for spider phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Performance on a Behavioral Approach Test in a Generalization Context (Pre-treatment to 2-week Follow-Up) | Change from pre-treatment (same day as treatment) to follow-up (window of 14-21 days after treatment)
  Change in peak subjective fear (0 - 100 scale), behavioral approach (0 - 13 scale), and physiological reactivity (heart rate and skin conductance) to a live spider not used during treatment (generalization context) from pre-treatment to follow-up

SECONDARY OUTCOMES:
Change in Performance on a Behavioral Approach Test in a Generalization Context (Pre-treatment to Post-treatment) | Change from pre-treatment (same day as treatment) to post-treatment (within 30 minutes of completion of the treatment procedure)
  Change in peak subjective fear (0 - 100 scale), behavioral approach (0 - 13 scale), and physiological reactivity (heart rate and skin conductance) to a live spider not used during treatment (generalization context) from pre-treatment to post-treatment.
Change in Performance on a Behavioral Approach Test in the Treatment Context (Pre-treatment to 2-week Follow-Up) | Change from pre-treatment (same day as treatment) to follow-up (window of 14-21 days after treatment)
  Change in peak subjective fear (0 - 100), behavioral approach (0 - 10), and physiological reactivity (heart rate and skin conductance) to a live spider used during treatment (treatment context) from pre-treatment to follow-up
Change in Performance on a Behavioral Approach Test in the Treatment Context (Pre-treatment to Post-treatment) | Change from pre-treatment (same day as treatment) to post-treatment (within 30 minutes of completion of the treatment procedure)
  Change in peak subjective fear (0 - 100), behavioral approach (0 - 10), and physiological reactivity (heart rate and skin conductance) to a live spider used during treatment (treatment context) from pre-treatment to post-treatment.
Change in Fear of Spiders Questionnaire (Pre-treatment to 2-week Follow-Up) | Change from pre-treatment (same day as treatment) to follow-up (window of 14-21 days after treatment)
  Change in psychometrically validated questionnaire assessing spider phobia severity from pre-treatment to follow-up.
Change in Armfield and Mattiske Disgust Questionnaire (Pre-treatment to 2-week Follow-Up) | Change from pre-treatment (same day as treatment) to follow-up (window of 14-21 days after treatment)
  Change in psychometrically validated questionnaire assessing severity of disgust response related to spider phobia from pre-treatment to follow-up.
Change in Spider Belief Questionnaire from pre-treatment to follow-up (Pre-treatment to 2-Week Follow-Up) | Change from pre-treatment (same day as treatment) to follow-up (window of 14-21 days after treatment)
  Change in psychometrically validated questionnaire assessing cognitions related to spider phobia from pre-treatment to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, PhD, Study Director — The University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No